CLINICAL TRIAL: NCT00251524
Title: A Phase II Study of Eloxatin and Alimta in Combination With Bevacizumab in Advanced Non-Squamous NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veeda Oncology (Other)
Collaborators: Sanofi (Industry); Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-04-015
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Oxaliplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab, Oxaliplatin, Pemetrexed — Avastin 15 mg/kg IV, Alimta 500 mg/m2 IV given over 10 minutes, Eloxatin 120 mg/m2 IV given over 2 hours
  Other Names: Avastin

SUMMARY:
This is a Phase II, open-label, non-randomized study in patients with advanced non-squamous NSCLC.

Each cycle will be 21 days. Patients will be evaluated every 2 cycles (~6 weeks) for response using RECIST criteria. Those patients achieving stable disease or better will continue therapy. Those patients experiencing progressive disease will be taken off study.

Patients will receive 6 cycles of Eloxatin, Alimta, and Bevacizumab. After the 6 cycles, patients will receive Bevacizumab alone every 21 days until evidence of disease progression or unacceptable toxicity.

Note: Once patient has completed the 6 cycles of Eloxatin, Alimta, and Bevacizumab and is receiving single-agent Bevacizumab, assessment of response will be performed every 3 cycles (~every 9 weeks) using RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must fulfill all of the following criteria:

* Patients or their legal representatives must be able to read and understand, and must have signed an IRB-approved informed consent to participate in the trial.
* Patients may have measurable or non-measurable disease based on RECIST criteria. Tumor lesions that are situated in a previously irradiated area are not considered measurable.
* Patients must have histologically documented Stage IIIB/IV non-squamous cell NSCLC.
* Patients must have an ECOG Performance Status of 0 or 1.
* Patients must be >18 years of age.
* Patients must either be not of child bearing potential or have a negative serum pregnancy test within 7 days prior to registration. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal for at least 12 months.
* Patients of childbearing potential must agree to use effective contraceptive measures during study treatment and for 90 days after receiving last study treatment.
* Patients must have white blood cell (WBC) >3,000/µL, absolute neutrophil count (ANC) >1,500/µL, platelets >100,000/µL, and hemoglobin >9g/dL.
* Calculated creatinine clearance (CrCl) <45mL/min based on the standard Cockroft and Gault formula.
* Patients must have a serum creatinine <1.5 x institutional upper limit of normal (ULN).
* Patients must have a bilirubin <1.5 x ULN, an ALT or AST <3 x ULN, and an alkaline phosphatase <3 x ULN. For patients with liver metastases, ALT, AST, and alkaline phosphatase levels can be <5 x ULN.
* Patients must have INR <1.5, and PTT <ULN within 1 week prior to registration.
* Urine Protein: Creatinine ratio must be < 1.0.

Exclusion Criteria:

Any of the following criteria will make the patient ineligible to participate in this study:

* Prior chemotherapy or biologic therapy, including prior treatment with Bevacizumab, for the treatment of non-squamous NSCLC.
* Patients with squamous cell NSCLC.
* Patients with any histology in close proximity to a major vessel, cavitation, or history of hemoptysis (bright red blood of 1/2 teaspoon or more).
* Patients who have a history of hypersensitivity to Eloxatin (or other platinum components), Alimta, or Bevacizumab or any of the components in these drugs.
* Patients who have undergone major surgery, open biopsy, or significant traumatic injury within 28 days prior to registration or anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to registration.
* Patients who received radiotherapy to more than 25% of their bone marrow; patients who received any radiotherapy within 4 weeks of registration, or previous radiation to the only area of measurable disease.
* Blood pressure of >150/100 mmHg, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (Appendix IV), or a history of myocardial infarction or stroke within 6 months.
* Clinically significant peripheral vascular disease or evidence of bleeding diathesis (prone to bleeding), or coagulopathy.
* Patients on therapeutic anticoagulation. (Prophylactic anticoagulation of venous access devices is allowed.)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of allogeneic transplant.
* Known HIV or Hepatitis B or C (active, previously treated, or both).
* Patients planning to receive any concurrent therapy to treat NSCLC during the study treatment period.
* Patients must not be receiving chronic daily treatment with Aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory agents known to prohibit platelet function. Treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix), or cilostazal (Pletal) is also not allowed.
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).
* Patients with a serious uncontrolled intercurrent medical or psychiatric illness, including an active infection, or a fever > 38.5°C within 3 days of the first scheduled day of study treatment.
* Patients with a history of other malignancy within the last 5 years, with the exception of low grade prostate cancer (Gleason Grades 1-4), non melanoma skin cancer, or carcinoma in situ of the cervix, which could affect the diagnosis or assessment of these study drugs for NSCLC. Patients treated more than 5 years ago for a malignancy other than non-squamous NSCLC are eligible.
* Patients with brain metastases or leptomeningeal disease.
* Any patient who is pregnant or lactating.
* Any patient who is unable to comply with requirements of study.
* Patients with peripheral neuropathy >grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine the median progression-free survival in patients with advanced non-squamous non-small cell lung cancer (NSCLC) receiving Eloxatin and Alimta in combination with Bevacizumab as first-line treatment | unk

SECONDARY OUTCOMES:
To evaluate the median and the 1-year and 2-year survival in patients with advanced NSCLC receiving Eloxatin and Alimta in combination with Bevacizumab as first-line treatment. | unk
To determine the overall objective response and the duration of response in patients with advanced NSCLC receiving Eloxatin and Alimta in combination with Bevacizumab as first-line treatment. | unk
To evaluate the safety of Eloxatin and Alimta in combination with Bevacizumab in patients with advanced NSCLC as first-line treatment. | unk

CONTACTS AND LOCATIONS:
Overall Officials: John Waples, MD, Principal Investigator — Veeda Oncology
Locations (1):
- Veeda Oncology, Columbus, Ohio, United States